CLINICAL TRIAL: NCT04136314
Title: The Effects of Gain- Versus Loss-Framed Messages on Patient Preferences for Therapies in Individuals With Psoriasis
Brief Title: Impact of Decision-Framing in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, April Armstrong, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS-19-00740
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Psoriasis Vulgaris; Psoriatic Arthritis; Psoriasis
Keywords: Decision-Framing; Prospect Theory; Medication Preferences
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Primary/blinded investigator will be blinded to randomization of subject to either group A (gain-framed) or group B (loss-framed) arms. Blinded party will create the randomization master list and provide a given subject's arm allocation to the primary/unblinded investigator once that subject has been enrolled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gain-Frame Survey [A] (Experimental)
  Interventions: Behavioral: Decision-Framed Survey
- Loss-Frame Survey [B] (Experimental)
  Interventions: Behavioral: Decision-Framed Survey

INTERVENTIONS:
Behavioral: Decision-Framed Survey — Survey will ask all subjects for will be asked to indicate basic demographic information, such as age, sex, race, and education level. Also, subjects will indicate whether they have been diagnosed with psoriatic arthritis. Importantly, patients will complete the survey questions anonymously, and no direct patient identifiers or HIPPA-protected information will be collected. Subjects will then be asked to indicate their preference for a hypothetical injectable medication after exposure to [A] a gain-framed message or [B] a loss-framed message.

SUMMARY:
Rationale:

Shared decision-making models between clinicians and patients are critical to improving healthcare delivery and adherence to medication. One type of model, decision framing, is rarely studied in medicine. Decision framing is the way that a choice is worded. In a clinical context, patient choices can be worded positively, or "gain-framed", to explain the benefits of a therapy or negatively, or "loss-framed", to explain the risks of not taking a therapy. Previous literature suggests that decision-framing can significantly influence patients' decision-making regarding their healthcare. However, a critical gap exists in understanding how decision framing affects psoriasis patients' preferences for therapies.

Objective:

Determine whether loss-framed messages lead to greater therapy acceptance as compared to gain-framed messages among adults with psoriasis.

Study population:

90 adults with psoriasis will be enrolled from USC ambulatory clinics and the general public.

Intervention:

Subjects will be exposed to gain-framed or loss-framed messages regarding psoriasis therapies. Specifically, gain-framed messages will explain the expected benefits of taking the psoriasis therapy and loss-framed messages will explain the potential risks of not taking the psoriasis therapy.

Study Methodology:

Cross-sectional single-intervention survey.

DETAILED DESCRIPTION:
Study Design:

The investigators will conduct a single intervention cross-sectional study to evaluate the impact of gain-framing versus loss-framing on patients' therapy preferences. This pragmatic study will compare whether patients are more likely to adhere to a hypothetical injectable psoriasis medication after exposure to a short paragraph explaining either the potential benefits after receiving the medication or the potential losses of not receiving the medication. The goal of this pragmatic study is to test whether differences arise in patient preferences depending on how the information they receive is framed.

Recruitment:

The investigators will recruit ninety adults with psoriasis from the Keck Medicine of University of Southern California (USC) Outpatient Care Network and the Los Angeles County+University of Southern California (LAC+USC) Medical Center outpatient clinic network.

Survey Administration:

Ninety subjects will be randomized using the HIPAA-compliant database Research Electronic Data Capture (REDCap) 1:1 to receive a survey regarding a hypothetical therapeutic intervention specific to their disease. All subjects (N=90) will be asked to indicate basic demographic information, such as age, sex, race, and education level. Also, the investigators will ask whether they have been diagnosed with psoriatic arthritis. Importantly, subjects will complete the survey questions anonymously, and no direct patient identifiers or HIPPA-protected information will be collected.

Half of the subjects (n=45) will be presented with a gain-framed message that explains the benefits of receiving a hypothetical injectable psoriasis medication. The other half (n=45) will be presented with a loss-framed message that explains the harms associated with not taking the medication. Both arms will include the same information regarding the possible side effects upon receiving the injection. The following are examples of gain-framed versus loss-framed messages for this study.

Example of a gain-framed question: A new injectable medication is being developed for psoriasis and psoriatic arthritis. If you take this medication, you will have the chance to reduce psoriasis severity, reduce joint pain, and improve how you feel overall. The side effects of this medication include a small chance of pain around the injection site and a small chance of skin infections. How likely are you to take this medication?

Example of a loss-framed question: A new injectable medication for psoriasis is being developed. If you do not take this medication, you will miss out on the chance to improve your skin, your joints, and your overall health. If you do not take this medication, your psoriasis may get worse; you may have worsening pain in your joints from psoriatic arthritis; and you may feel worse overall. The side effects of this medication include a small chance of pain around the injection site and a small chance of skin infections. How likely are you to take this medication?

After each arm is exposed to their respective gain-framed or loss-framed question, each participant will be asked to indicate their preference on a scale from zero to ten. Zero indicates they definitely will not use the medication while ten indicates they definitely will use the medication.

The investigators will not collect any patient protected information, such as name, date of birth, phone numbers, or address. Subjects will fill out the survey anonymously.

Selection of Participants:

With a total sample size of 90 (45 per each group), this study has 80% power to detect a difference of 1.5 in the means between the subjects randomized to positively framed messages versus those randomized to negative framed messages with alpha of 0.05 and standard deviation of 2.5.

Statistical Analysis: The investigators will perform a multivariate regression analysis and a paired t-test to determine statistical and clinical significance. To minimize confounding, the multivariate regression analysis will adjust for demographic and clinical characteristics such as gender and the presence or absence of psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Has physician diagnosed psoriasis with or without psoriatic arthritis
* Able to read and write in either English or Spanish

Exclusion Criteria:

* Less than 18 years of age
* Does not have physician diagnosed psoriasis
* Unable to read and respond to questionnaires in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Gain-framed vs. Loss-framed Survey Responses | Up to 14 weeks
  Difference in survey responses based on exposure to gain-frame or loss-frame question. After exposure to the positively or negatively framed question, subjects will be asked how likely they would agree to receive a hypothetical injectable medication. The subjects will answer with a Likert scale ranging from 0 to 10, with 0 indicating they will definitely not want the medication and 10 indicating they will definitely want the medication. Each enrolled subject will complete the survey only once.

SECONDARY OUTCOMES:
Effect of Psoriatic Arthritis on Survey Responses | Up to 14 weeks
  Difference in survey responses based on history of psoriatic arthritis. All study participants will be asked to include basic demographic information, such as their age, race, ethnicity, sex, and highest level of education. All subjects will also be asked whether they have ever been diagnosed with psoriatic arthritis. The investigators will then determine if stratifying the presence or absence of psoriatic arthritis impacts the subjects' response on the 11-point Likert scale described above.
Effect of Sex on Survey Responses | Up to 14 weeks
  Difference in survey responses based on subject sex. All study participants will be asked to include basic demographic information, such as their age, race, ethnicity, sex, and highest level of education. The investigators will then determine if stratification based on sex impacts the subjects' responses on the 11-point Likert scale described above.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States